CLINICAL TRIAL: NCT03589612
Title: Regression of Hamstring Flexibility and Performance in Children With Duchenne Muscular Dystrophy
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Lütfiye AKKURT, PT, Principal investigator, Hacettepe University
Other Study IDs: GO 16/740-2
Record Dates: First submitted 2018-07-05; First posted 2018-07-18 (Actual); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: Duchenne Muscular Dystrophy; Performance; Flexibility
Keywords: Duchenne Muscular Dystrophy; performance; hamstring flexibility; regression
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Investigator investigated that regression of hamstring flexibility and performance in children with Duchenne Muscular Dystrophy.

DETAILED DESCRIPTION:
Flexibility of hamstrings was evaluated by Popliteal Angle test. Performance was evaluated 6 Minute Walk Test (6 MWT). Regression of hamstring flexibility and performance was examined regression tests. Correlation was examined between popliteal angle test and parameter of North Star Ambulation Assessment.

ELIGIBILITY:
Inclusion Criteria:

* To be a Duchenne Muscular Dystrophy diagnosis,
* Being in the ambulatory period and climbing four steps independently,
* to be Level 1 and Level 2 according to Brooke Lower Functional Classification Test
* To be able to cooperate
* No any severe contracture in the lower limbs which may prevent assessments,

Exclusion Criteria:

* Children who fail to meet these criteria study.

Ages: 5 Years to 14 Years | Sex: Male
Age Groups: Child
Study Population: Sixty children will participated this study. Fourty-two children was assessed, and eighteen children will assess in a few months.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2018-03-08 (Actual); Primary Completion 2019-01-24 (Actual); Study Completion 2019-01-24 (Actual)

PRIMARY OUTCOMES:
Popliteal Angle Test | 5 minute
  The Popliteal Angle Test was used to assess hamstring flexibility. Child asked to rise lower leg straight. Incomplete angle degree of full extension is popliteal angle.

SECONDARY OUTCOMES:
6 Minute Walk Test | 6 minute
  6 Minute Walk Test was used to assess performance with children Duchenne MUscular Dystropy.
North Star Ambulation Assessment | 20 minute
  The North Star Ambulatory Assessment (NSAA) is used to assess mobility for in ambulatory children with DMD for 5 years. NSAA is consist of 17 items from stand to run.

CONTACTS AND LOCATIONS:
Overall Officials: Güllü Aydın, Msc., Principal Investigator — Hacettepe University; Numan Bulut, Msc, Principal Investigator — Hacettepe University; İpek Gürbüz, Assoc.Prof., Principal Investigator — Hacettepe University; Ayşe Karaduman, Prof., Principal Investigator — Hacettepe University; Oznur Yılmaz, Study Director — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Sıhhiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No